CLINICAL TRIAL: NCT02525900
Title: Comparing the Efficacy of Transversus Abdominis Plane Block, Both Single Injection and Continuous Block Technique, to Wound Infiltration for Total Abdominal Hysterectomy: A Prospective Randomized Study
Brief Title: ssTAP vs TAP Catheters in TAH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow enrollment, and unusable data
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204411
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wound Infiltration (Placebo Comparator): 0.5mg/kg of 0.25% bupivacaine will be injected around the incision for wound infiltration
  Interventions: Procedure: Wound Infiltration
- TAP Blocks (Experimental): 20mL of 0.25% bupivacaine will be injected on each side of the abdomen for ssTAP procedures
  Interventions: Procedure: TAP Blocks
- TAP Catheters (Experimental): 20mL of 0.25% bupivacaine will be injection on each side of the abdomen and catheters placed for repeat bolus every 12 hours with 20mL of 0.25% Bupivacine until 48 hours post procedure or hospital discharge.
  Interventions: Procedure: TAP Catheters

INTERVENTIONS:
Procedure: Wound Infiltration — Wound Infiltration with 0.25% Bupivacine
  Arms: Wound Infiltration
Procedure: TAP Blocks — bilateral TAP block with 0.25% Bupivacaine
  Arms: TAP Blocks
Procedure: TAP Catheters — bilateral TAP Catheter with repeat bolus of 0.25% Bupivacaine
  Arms: TAP Catheters

SUMMARY:
Prospective, randomized study comparing local wound infiltration with local anesthetic (LA) versus single injection TAP blocks (ssTAP) with LA versus continuous TAP block (TAP caths) catheters with LA for treatment of postoperative pain after total abdominal hysterectomy (TAH).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo total abdominal hysterectomy
* Age ≥ 18 years.
* American Society of Anesthesiologists (ASA) physical status ≤ 3

Exclusion Criteria:

* Known coagulopathy
* Known allergy to Bupivacaine or morphine
* Contraindication to Tylenol usage
* Medical conditions contraindicated to bupivacaine use
* Daily narcotic usage for ≥ 2 weeks of 20mg of oxycodone daily or an equivalent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption postoperatively for pain management as measured by the Visual Analog Scale (VAS) pain scale. | Up to 48 hours post treatment
  The total morphine consumption used post operatively to manage pain will be measured utilizing the VAS pain scale with 0 being no pain and 10 being as much pain as can be tolerated.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tingle, M.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided